CLINICAL TRIAL: NCT01502657
Title: Ultrasound Guided Percutaneous Tracheostomy in the ICU
Brief Title: Ultrasound Guided Percutaneous Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PI10-DR-GUINOT; 2010-A00901-38 (Other: RCB)
Record Dates: First submitted 2011-04-21; First posted 2012-01-02 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Tracheostomy Hemorrhage; Tracheostomy Complications; Other Tracheostomy Complications
Keywords: percutaneous tracheostomy; ultrasonography; echography; critical care
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultrasonography (EnVisor Philips Medical Systems) — Percutaneous tracheostomy is performed using the dilatational method with ultrasonography guidance;
  Other Names: Echograph is EnVisor Philips; N°453561299512 rev A; CE0086

SUMMARY:
The purpose of this study is to determine the feasibility and the safety of ultrasound guided percutaneous dilatational tracheostomy.

DETAILED DESCRIPTION:
Percutaneous tracheostomy is commonly performed in critical care units when ventilatory weaning fails or when prolonged mechanical ventilation is required. Numerous complications have been described since the widespread use of Percutaneous Tracheostomy (PCT). Bronchoscopy-guided percutaneous tracheostomy was developed in this context. However, bronchoscopy cannot identify vascular structures and the thyroid gland in the neck, and therefore cannot prevent complications related to organ lesions in the neck. Several studies have demonstrated the value of ultrasound guidance in the neck before performing PCT. No studies have demonstrated the feasibility and the safety of ultrasound guidance for PCT. Ultrasound could improve the understanding of neck anatomy, prevents vascular puncture, and helps guide insertion of the tracheostomy tube.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in ICU in whom percutaneous tracheostomy is indicated,
* patients aged > 18 years old,

Exclusion Criteria:

* age less than 18 years,
* clotting disorder,
* infection at the puncture site,
* emergency tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Procedure related complications | At the end of the procedure, then participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Complications are: paratracheal insertion, injuries to blood vessels in the neck, oesophageal injury, accidental decannulation, malposition of the tracheostomy tube, tracheal cuff puncture, multiple punctures (more than 3), surgical conversion and percutaneous tracheostomy failure, bleeding (compressible, incompressible, requiring administration of labile blood products), pneumothorax, pneumomediastinum, tracheostomy puncture site infection, surgical conversion, subglottic stenosis, fracture of a tracheal cartilage, granuloma.

SECONDARY OUTCOMES:
Procedure time | The time will be calculated at the end of the procedure; an average of 30 minutes
  The total time consisted of a first phase of ulstrasound examination of the cervical region and an implementation phase under ultrasound of percutaneous tracheostomy.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre grégoire Guinot, MD, Principal Investigator — Centre Hospitalier Universitaire, Amiens
Locations (1):
- CHU Amiens, Amiens, Somme, France

REFERENCES:
- [Result] Guinot PG, Zogheib E, Petiot S, Marienne JP, Guerin AM, Monet P, Zaatar R, Dupont H. Ultrasound-guided percutaneous tracheostomy in critically ill obese patients. Crit Care. 2012 Dec 12;16(2):R40. doi: 10.1186/cc11233. PMID 22390815